CLINICAL TRIAL: NCT00502320
Title: Randomized Placebo-Controlled Trial of Ramelteon in the Treatment of Sleep and Mood in Patients With Seasonal Affective Disorder
Brief Title: Ramelteon in the Treatment of Sleep and Mood in Patients With Seasonal Affective Disorder
Acronym: SAM-SAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lehigh Valley Hospital (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Edward R. Norris, MD, Lehigh Valley Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06-006R
Record Dates: First submitted 2007-07-13; First posted 2007-07-17 (Estimated); Results first posted 2009-10-05 (Estimated); Last update posted 2009-10-06 (Estimated); Status verified 2009-10

CONDITIONS: Seasonal Affective Disorder
Keywords: Seasonal Affective Disorder; Ramelteon; Psychiatry; Randomized Controlled Trial; Hamilton Depression Rating Scale- SAD Version; Circadian Rhythm
MeSH Terms: conditions — Seasonal Affective Disorder | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ramelteon (Experimental): 8 mg
  Interventions: Drug: Ramelteon
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ramelteon — one 8 mg tablet at bed for up to 4 months
  Other Names: Rozerem
  Arms: Ramelteon
Drug: Placebo — one tablet at bedtime for up to 4 months
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether treating sleep difficulties in patients with seasonal affective disorder also improves their depressive symptoms.

DETAILED DESCRIPTION:
Seasonal affective disorder(SAD) is a type of depression in which a patient's depressive symptoms worsen in the winter. These patients' depressive symptoms often lessen in the spring and summer months. Much of the focus of the treatment of SAD (light therapy and melatonin) has involved the brain's suprachiasmatic nucleus(SCN), as it is hypothesized that one potential reason for SAD is a desynchronized SCN. Ramelteon offers a new and more pharmacologically exact mechanism to re-synchronize the SCN. The administration of ramelteon for this patient population may improve sleep, and in addition, do so in a manner that may also reduce their seasonal affective depressive symptoms. Patients eligible for enrollment will be administered either ramelteon or placebo and return to the study office for 4 monthly visits over the winter months, to evaluate the effects of ramelteon versus placebo on sleep and mood.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18-65 yrs.
* A diagnosis of seasonal affective disorder
* A Pittsburgh Sleep Quality Index >5
* English speaking
* Be able to sign informed consent

Exclusion Criteria:

* Active substance abuse
* Current psychotic symptoms
* Severe personality disorders
* Primary sleep disorders
* Severe chronic obstructive pulmonary disease (COPD)
* Prescription fluvoxamine(Luvox) use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-09; Primary Completion 2008-04 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward R. Norris, MD, Principal Investigator — Lehigh Valley Hospital
Locations (1):
- Lehigh Valley Hospital, Department of Psychiatry, Allentown, Pennsylvania, United States

REFERENCES:
- [Background] Avery DH, Eder DN, Bolte MA, Hellekson CJ, Dunner DL, Vitiello MV, Prinz PN. Dawn simulation and bright light in the treatment of SAD: a controlled study. Biol Psychiatry. 2001 Aug 1;50(3):205-16. doi: 10.1016/s0006-3223(01)01200-8. PMID 11513820
- [Background] Biggs JT, Wylie LT, Ziegler VE. Validity of the Zung Self-rating Depression Scale. Br J Psychiatry. 1978 Apr;132:381-5. doi: 10.1192/bjp.132.4.381. PMID 638392
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Hoch CC, Yeager AL, Kupfer DJ. Quantification of subjective sleep quality in healthy elderly men and women using the Pittsburgh Sleep Quality Index (PSQI). Sleep. 1991 Aug;14(4):331-8. PMID 1947597
- [Background] Desan PH, Weinstein AJ, Michalak EE, Tam EM, Meesters Y, Ruiter MJ, Horn E, Telner J, Iskandar H, Boivin DB, Lam RW. A controlled trial of the Litebook light-emitting diode (LED) light therapy device for treatment of Seasonal Affective Disorder (SAD). BMC Psychiatry. 2007 Aug 7;7:38. doi: 10.1186/1471-244X-7-38. PMID 17683643
- [Background] Dubocovich ML, Rivera-Bermudez MA, Gerdin MJ, Masana MI. Molecular pharmacology, regulation and function of mammalian melatonin receptors. Front Biosci. 2003 Sep 1;8:d1093-108. doi: 10.2741/1089. PMID 12957828
- [Background] Gentili A, Weiner DK, Kuchibhatla M, Edinger JD. Test-retest reliability of the Pittsburgh sleep quality index in nursing home residents. J Am Geriatr Soc. 1995 Nov;43(11):1317-8. doi: 10.1111/j.1532-5415.1995.tb07415.x. No abstract available. PMID 7594173
- [Background] Golden RN, Gaynes BN, Ekstrom RD, Hamer RM, Jacobsen FM, Suppes T, Wisner KL, Nemeroff CB. The efficacy of light therapy in the treatment of mood disorders: a review and meta-analysis of the evidence. Am J Psychiatry. 2005 Apr;162(4):656-62. doi: 10.1176/appi.ajp.162.4.656. PMID 15800134
- [Background] Hellpach, W.H. (1911). Die geopsychischen erschelnungen; Wetter und klima und landschaft in ihrem einfluss auf das seelenleben. Leipzig: W. Engelmann.
- [Background] Jenner FA. Chronobiology and the clinical psychiatrist: the current position. Chronobiologia. 1974 Apr-Jun;1(2):151-60. No abstract available. PMID 4617659
- [Background] Lam RW, Gorman CP, Michalon M, Steiner M, Levitt AJ, Corral MR, Watson GD, Morehouse RL, Tam W, Joffe RT. Multicenter, placebo-controlled study of fluoxetine in seasonal affective disorder. Am J Psychiatry. 1995 Dec;152(12):1765-70. doi: 10.1176/ajp.152.12.1765. PMID 8526243
- [Background] Levitt AJ, Lam RW, Levitan R. A comparison of open treatment of seasonal major and minor depression with light therapy. J Affect Disord. 2002 Sep;71(1-3):243-8. doi: 10.1016/s0165-0327(01)00397-4. PMID 12167524
- [Background] Lewy AJ, Sack RL. The phase-shift hypothesis of seasonal affective disorder. Am J Psychiatry. 1988 Aug;145(8):1041-3. doi: 10.1176/ajp.145.8.1041c. No abstract available. PMID 3394867
- [Background] Lewy AJ, Lefler BJ, Emens JS, Bauer VK. The circadian basis of winter depression. Proc Natl Acad Sci U S A. 2006 May 9;103(19):7414-9. doi: 10.1073/pnas.0602425103. Epub 2006 Apr 28. PMID 16648247
- [Background] Liu C, Weaver DR, Jin X, Shearman LP, Pieschl RL, Gribkoff VK, Reppert SM. Molecular dissection of two distinct actions of melatonin on the suprachiasmatic circadian clock. Neuron. 1997 Jul;19(1):91-102. doi: 10.1016/s0896-6273(00)80350-5. PMID 9247266
- [Background] Manber R, Blasey C, Arnow B, Markowitz JC, Thase ME, Rush AJ, Dowling F, Koscis J, Trivedi M, Keller MB. Assessing insomnia severity in depression: comparison of depression rating scales and sleep diaries. J Psychiatr Res. 2005 Sep;39(5):481-8. doi: 10.1016/j.jpsychires.2004.12.003. Epub 2005 Jan 23. PMID 15992557
- [Background] McClung CA. Circadian genes, rhythms and the biology of mood disorders. Pharmacol Ther. 2007 May;114(2):222-32. doi: 10.1016/j.pharmthera.2007.02.003. Epub 2007 Feb 28. PMID 17395264
- [Background] Michalak EE, Wilkinson C, Dowrick C, Wilkinson G. Seasonal affective disorder: prevalence, detection and current treatment in North Wales. Br J Psychiatry. 2001 Jul;179:31-4. doi: 10.1192/bjp.179.1.31. PMID 11435265
- [Background] Michalak EE, Murray G, Levitt AJ, Levitan RD, Enns MW, Morehouse R, Tam EM, Cheung A, Lam RW. Quality of life as an outcome indicator in patients with seasonal affective disorder: results from the Can-SAD study. Psychol Med. 2007 May;37(5):727-36. doi: 10.1017/S0033291706009378. Epub 2006 Nov 20. PMID 17112403
- [Background] Modell JG, Rosenthal NE, Harriett AE, Krishen A, Asgharian A, Foster VJ, Metz A, Rockett CB, Wightman DS. Seasonal affective disorder and its prevention by anticipatory treatment with bupropion XL. Biol Psychiatry. 2005 Oct 15;58(8):658-67. doi: 10.1016/j.biopsych.2005.07.021. PMID 16271314
- [Background] Moscovitch A, Blashko CA, Eagles JM, Darcourt G, Thompson C, Kasper S, Lane RM; International Collaborative Group on Sertraline in the Treatment of Outpatients with Seasonal Affective Disorders. A placebo-controlled study of sertraline in the treatment of outpatients with seasonal affective disorder. Psychopharmacology (Berl). 2004 Feb;171(4):390-7. doi: 10.1007/s00213-003-1594-8. Epub 2003 Sep 19. PMID 14504682
- [Background] Pjrek E, Winkler D, Kasper S. Pharmacotherapy of seasonal affective disorder. CNS Spectr. 2005 Aug;10(8):664-9; quiz 672. doi: 10.1017/s1092852900019623. PMID 16041297
- [Background] Postolache TT, Oren DA. Circadian phase shifting, alerting, and antidepressant effects of bright light treatment. Clin Sports Med. 2005 Apr;24(2):381-413, xii. doi: 10.1016/j.csm.2004.12.005. PMID 15892931
- [Background] Praschak-Rieder N, Willeit M, Wilson AA, Houle S, Meyer JH. Seasonal variation in human brain serotonin transporter binding. Arch Gen Psychiatry. 2008 Sep;65(9):1072-8. doi: 10.1001/archpsyc.65.9.1072. PMID 18762593
- [Background] Rohan KJ, Roecklein KA, Tierney Lindsey K, Johnson LG, Lippy RD, Lacy TJ, Barton FB. A randomized controlled trial of cognitive-behavioral therapy, light therapy, and their combination for seasonal affective disorder. J Consult Clin Psychol. 2007 Jun;75(3):489-500. doi: 10.1037/0022-006X.75.3.489. PMID 17563165
- [Background] Rosenthal NE, Sack DA, Gillin JC, Lewy AJ, Goodwin FK, Davenport Y, Mueller PS, Newsome DA, Wehr TA. Seasonal affective disorder. A description of the syndrome and preliminary findings with light therapy. Arch Gen Psychiatry. 1984 Jan;41(1):72-80. doi: 10.1001/archpsyc.1984.01790120076010. PMID 6581756
- [Background] Ruhrmann S, Kasper S, Hawellek B, Martinez B, Hoflich G, Nickelsen T, Moller HJ. Effects of fluoxetine versus bright light in the treatment of seasonal affective disorder. Psychol Med. 1998 Jul;28(4):923-33. doi: 10.1017/s0033291798006813. PMID 9723147
- [Background] Thompson, C. (2001). Evidence-based treatment. In Seasonal Affective Disorder: Practice and Research (ed. T. Partonen and A. Magnusson), 151-158. New York: Oxford University Press.
- [Background] Thurber S, Snow M, Honts CR. The Zung Self-Rating Depression Scale: convergent validity and diagnostic discrimination. Assessment. 2002 Dec;9(4):401-5. doi: 10.1177/1073191102238471. PMID 12462760
- [Background] Willeit M, Praschak-Rieder N, Neumeister A, Zill P, Leisch F, Stastny J, Hilger E, Thierry N, Konstantinidis A, Winkler D, Fuchs K, Sieghart W, Aschauer H, Ackenheil M, Bondy B, Kasper S. A polymorphism (5-HTTLPR) in the serotonin transporter promoter gene is associated with DSM-IV depression subtypes in seasonal affective disorder. Mol Psychiatry. 2003 Nov;8(11):942-6. doi: 10.1038/sj.mp.4001392. PMID 14593433
- [Background] William JBW, Link MJ, Rosenthal NE, Terman M. (1988). Structured Interview Guide for the Hamilton Depression Rating Scale, Seasonal Affective Disorders Version (SIGH-SAD). New York, New York State Psychiatric Institute
- [Background] ZUNG WW. A SELF-RATING DEPRESSION SCALE. Arch Gen Psychiatry. 1965 Jan;12:63-70. doi: 10.1001/archpsyc.1965.01720310065008. No abstract available. PMID 14221692
- [Background] Zung WW. Factors influencing the self-rating depression scale. Arch Gen Psychiatry. 1967 May;16(5):543-7. doi: 10.1001/archpsyc.1967.01730230027003. No abstract available. PMID 4381571
- [Background] American Psychiatric Association: Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision. Washington, DC, American Psychiatric Association, 2000.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in August 2006 and was completed by October 2007. Participants, who at the time were receiving outpatient psychiatric services through Lehigh Valley Hospital, were recruited via referral through the department of psychiatry, and also through print advertisement. Participants received no compensation for participating in the study.
Pre-assignment Details: 50 individuals signed the informed consent document, one was a screen failure, so 49 participants started study medication. During the study, both treatment groups were maintained on their usual medications for depression and allowed treatment as usual, including medication adjustments.
Groups:
- Ramelteon: 8 mg pill taken by mouth nightly
- Placebo: inactive sugar pill taken by mouth nightly
Period: Overall Study
Arm/Group | Ramelteon | Placebo
Started | 25 | 25
Screening Visit | 25 | 24 (Participant signed informed consent but was a screen failure because she was nursing at the time.)
Completed | 19 | 18
Not Completed | 6 | 7
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrew Consent | 1 | 0
Not completed — No longer met criteria | 1 | 0
Not completed — Screen Failure | 0 | 1
Not completed — Adverse Event | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ramelteon | Placebo | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 45.49 (11.81) | 47.76 (10.23) | 46.08 (11.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 6 | 7 | 13
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Sleep Satisfaction at Baseline and Measured Monthly, as Measured by the Pittsburgh Sleep Quality Index (PSQI)
Description: Self-rated scale to measure quality of sleep via questions regarding sleep latency, duration, efficiency, disturbances, use of sleep medication, and daytime dysfunction. Score ranges from 0-21, higher scores represent more significant sleep disturbance.
Time Frame: Monthly for duration of treatment (up to 4 months)
Population: Intention to Treat analysis; excludes one screen failure.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 25 | 24
scores on a scale
  Baseline | 11.56 (0.75) | 11.45 (0.77)
  Month 1 | 9.52 (0.84) | 8.67 (0.90)
  Month 2 | 7.57 (0.84) | 8.62 (0.89)
  Month 3 | 8.07 (0.83) | 9.88 (0.85)
  Month 4 | 7.05 (0.85) | 9.61 (0.87)

2. Secondary Outcome: Depressive Symptoms at Baseline and Measured Monthly, as Measured by the Zung Depression Scale (ZDS)
Description: Self-rated scale to measure severity of depressive symptoms. Score ranges from 25-100, higher scores reflect more depression.
Time Frame: Monthly for duration of treatment (up to 4 months)
Population: Intention to Treat analysis; excludes one screen failure.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 25 | 24
scores on a scale
  Baseline | 63.06 (1.92) | 58.63 (1.96)
  Month 1 | 54.35 (2.70) | 56.40 (2.86)
  Month 2 | 53.51 (2.71) | 58.59 (2.80)
  Month 3 | 49.26 (2.81) | 58.62 (2.89)
  Month 4 | 46.14 (2.65) | 61.65 (2.74)

3. Secondary Outcome: Depressive Symptoms at Baseline and Measured Monthly, as Measured by the Structured Interview Guide for the Hamilton Depression Rating - Seasonal Affective Disorder (SIGH-SAD)
Description: Clinician-rated measure of mood; evaluates classical 21 Hamilton Depression items, and 8-item subscale measuring atypical depression symptoms which commonly occur during SAD episodes. Score ranges from 0-89, higher scores indicate higher levels of depression.
Time Frame: Monthly for duration of treatment (up to 4 months)
Population: Intention to Treat analysis; excludes one screen failure.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 25 | 24
scores on a scale
  Baseline | 22.68 (1.60) | 19.99 (1.63)
  Month 1 | 16.16 (1.88) | 15.97 (2.04)
  Month 2 | 14.81 (1.90) | 19.47 (1.96)
  Month 3 | 11.69 (1.66) | 20.65 (1.67)
  Month 4 | 9.15 (1.67) | 23.68 (1.71)

ADVERSE EVENTS:
Arm/Group | Ramelteon | Placebo
Serious Adverse Events (participants affected / at risk) | 1 | 0
Other Adverse Events (participants affected / at risk) | 2 | 5
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Ramelteon | Placebo
Worsening depression leading to hospitalization (Psychiatric disorders) | 1/25 (1) | 0/24 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Ramelteon | Placebo
Anxiety (Psychiatric disorders) | 1/25 (1) | 0/24 (0)
Depression (Psychiatric disorders) | 1/25 (1) | 1/24 (1)
Fatigue (General disorders) | 1/25 (1) | 1/24 (1)
Insomnia Exacerbation (General disorders) | 1/25 (1) | 3/24 (3)
Nightmares (General disorders) | 1/25 (1) | 0/24 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes